CLINICAL TRIAL: NCT01133431
Title: Clinical Study to Assess the Pharmacokinetic Interaction Between CKD-501 and Sulfonylurea (Glimepiride) in Healthy Male Subjects: Single-blinded, Randomized, Crossover Study
Brief Title: The Pharmacokinetic Interaction Between CKD-501 and Sulfonylurea
Acronym: CKD-501 DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Chong Kun Dang Pharmaceutical, Chong Kun Dang Pharmaceutical
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: CKD-19HPS10A
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-05

CONDITIONS: Healthy Male Volunteer
Keywords: CKD-501; Glimepiride; Placebo; Healthy male volunteer; Pharmacokinetic; Metabolite
MeSH Terms: interventions — lobeglitazone; Tablets; glimepiride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD-501 + Glimepiride -> CKD-501 placebo + Glimepiride (Experimental): This study is randomized, single-blinded, two-period, 2 treatments, crossover design to assess the pharmacokinetics interaction between CKD-501 and sulfonylurea.
  Interventions: Drug: CKD-501 0.5 mg tablet, Glimepiride 4 mg tablet; Drug: CKD-501 placebo tablet, Glimepiride 4 mg tablet
- CKD-501 placebo + Glimepiride -> CKD-501 + Glimepiride (Experimental): This study is randomized, single-blinded, two-period, 2 treatments, crossover design to assess the pharmacokinetics interaction between CKD-501 and sulfonylurea.
  Interventions: Drug: CKD-501 0.5 mg tablet, Glimepiride 4 mg tablet; Drug: CKD-501 placebo tablet, Glimepiride 4 mg tablet

INTERVENTIONS:
Drug: CKD-501 0.5 mg tablet, Glimepiride 4 mg tablet — From day 1 to day 4, CKD-501 0.5mg is administered daily to Group 1 patients during period 1. Then on day 5,CKD-501 0.5mg and glimepiride 4mg is co-administered to overnight-fasting Group 1 patients at period 1. After 10 day-break, period 2 will be repeated with CKD-501 placebo and glimepiride 4mg in Group 1.
  Other Names: CKD-501 : Lobeglitazone
Drug: CKD-501 placebo tablet, Glimepiride 4 mg tablet — From day 1 to day 4, CKD-501 placebo is administered daily to Group 2 patients during period 1. Then on day 5,CKD-501 placebo and glimepiride 4mg is co-administered to overnight-fasting Group 2 patients at period 1. After 10 day-break, period 2 will be repeated with CKD-501 0.5mg and glimepiride 4mg in Group 2.
  Other Names: CKD-501 : Lobeglitazone

SUMMARY:
To assess the pharmacokinetic Interaction between CKD-501 and sulfonylurea (Glimepiride) in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults aged between 20 and 45 during screening period
* Weight more than 45kg and within ±20% range of Ideal Boby Weight
* Agreement with written informed consent

Exclusion Criteria:

* Subject has signs of symptoms of acute disease within 28 days of starting administration of investigational drug
* Subject has a history(such as inflammatory gastrointestinal disease, gastric or duodenal ulcer, liver diseases, gastrointestinal surgical histories except for an appendectomy) affects the ADME of drug
* Clinically significant, active gastrointestinal system, cardiovascular system, pulmonary system, renal system, endocrine system, blood system, digestive system, central nervous system, mental disease or malignancy
* Inadequate subject by medical examination(medical history, physical examination, ECG, laboratory test) within 28 days of starting administration of investigational drug
* Inadequate laboratory test result

  * AST(SGOT) or ALT(SGPT) > 1.25 x upper limit of normal range
  * Total bilirubin > 1.5 x upper limit of normal range
* Clinically significant allergic disease(except for mild allergic rhinitis is not needed medication)
* Subject with known for hypersensitivity reactions to glitazones or sulfonylureas
* Previously participated in other trial within 60 days
* Medication with drug-mediated induction/inhibition metabolic enzyme such as barbiturates within 1 month or with may affect the clinical trial within 10 days
* Subject has taken abnormal meals which affects the ADME of drug
* Impossible to taking the institutional standard meal
* Previously donate whole blood within 60 days or component blood within 20 days
* Continued to be taking caffeine (caffeine > 5 cup/day), drinking(alcohol > 30 g/day) or cannot stop drinking or severe heavy smoker(cigarette > 10 cigarettes per day)during clinical trials
* An impossible one who participates in clinical trial by investigator's decision including laboratory test result

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the Pharmacokinetic Interaction between CKD-501 and sulfonylurea (Glimepiride) in healthy male subjects | 0-24 hrs
  Blood sampling timepoint : Day 1(0hr), Day 4(0hr), Day 5(0hr),0.5hr, 1hr, 1.5hr, 2hr, 2.5hr, 3hr, 3.5hr, 4hr, 5hr, 6hr, 8hr, 12hr, 24hr(Day 6)- total 16 timepoints per period

SECONDARY OUTCOMES:
To confirm and evaluate the pharmacokinetic characters of main metabolites of CKD-501 | 0-24 hrs
  Blood sampling timepoint : Day 1(0hr), Day 4(0hr), Day 5(0hr),0.5hr, 1hr, 1.5hr, 2hr, 2.5hr, 3hr, 3.5hr, 4hr, 5hr, 6hr, 8hr, 12hr, 24hr(Day 6)- total 16 timepoints per period

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Park, Ph.D., Principal Investigator — Korea University Anam Hospital
Locations (1):
- The Korea University Anam Hospital, Seoul, South Korea